CLINICAL TRIAL: NCT07011589
Title: Targeting Collagen VII Antibodies in Bullous Diseases Using Efgartigimod IV (VYVGART)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M. Peter Marinkovich (Other)
Collaborators: argenx (Industry)
Responsible Party: Sponsor-Investigator, M. Peter Marinkovich, Associate Professor of Dermatology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 74784
Record Dates: First submitted 2025-06-05; First posted 2025-06-09 (Actual); Last update posted 2025-06-09 (Actual); Status verified 2025-06

CONDITIONS: Epidermolysis Bullosa (EB); Epidermolysis Bullosa Acquisita; Recessive Dystrophic Epidermolysis Bullosa; Dystrophic Epidermolysis Bullosa
Keywords: epidermolysis bullosa; epidermolysis bullosa acquisita; dystrophic epidermolysis bullosa; recessive dystrophic epidermolysis bullosa; recessive; dystrophic; epidermolysis; bullosa; acquisita; collagven 7; c7; Col7; EB; EBA; DEB; RDEB; antibodies; Collagen VII; VII; IV IgG; IgG; IV; IVIgG; C7 antibodies; Collagen 7 antibodies; Collagen VII Antibodies; Vyjuvek; B-VEC; Efgartigimod
MeSH Terms: conditions — Epidermolysis Bullosa; Epidermolysis Bullosa Acquisita; Epidermolysis Bullosa Dystrophica | interventions — efgartigimod alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Efgartigimod (Experimental): There is one arm of the study. First, each participant undergoes a 3-month observational period. If the participant has DEB, they will continue their standard of care VYJUVEK as prescribed. After the observational period concludes, the participant enters the treatment period, during which Efgartigimod is administered. DEB participants will continue their standard of care VYJUVEK as prescribed.
  Interventions: Biological: Efgartigimod

INTERVENTIONS:
Biological: Efgartigimod — Dosage: 10mg/kg Frequency: Once a week Duration: 25 weeks
  Other Names: efgartigimod alfa; efgartigimod alfa fcab; VYVGART

SUMMARY:
The study objective is to see if IV Efgartigimod and Vyjuvek treatment in Recessive Dystrophic Epidermolysis Bullosa (RDEB) and IV Efgartigimod treatment in Epidermolysis Bullosa Acquisita (EBA) improves wound healing and affects the levels of C7 antibody levels in serum.

Fewer wounds, more rapidly healing wounds, and decreased C7 antibodies could improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* For DEB patients (aged 12 years or older): DEB confirmed with mutation analysis and correlated by phenotype, and treatment of at least 1 wound treated with topical gene therapy (VYJUVEK). Presence of C7 antibodies above normal cutoff on ELISA.
* For (classic) EBA patients (aged 18 years or older): EBA confirmed with positive histopathology (DIF), C7 antibodies above normal cutoff on ELISA, and having at least 1 skin lesion.
* The participant has a Karnofsky performance status of at least 60% at screening.
* Contraceptive use by reproductive male and female patients should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies and:

  1. Male participants:

     - Must agree to use an acceptable method of contraception and not donate sperm from the time that the ICF is signed until they have received their last dose of IMP.
  2. Female participants:

     * Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at week 1 / baseline before study intervention can be administered. Subsequent urine pregnancy tests are to be completed at week 6, week 11, week 16, week 21, and week 26 / EoS.
     * WOCBP must agree to use a highly effective or acceptable contraception method until at least 90 days after they receive their last dose of IMP.

Exclusion Criteria:

* Linear IgA dermatosis-like EBA or other autoimmune blistering diseases (including but not limited to pemphigus vulgaris, bullous pemphigoid, mucous membrane pemphigoid).
* Use of the following EBA treatments:

  * sulfasalazine, IVIg, subcutaneous administration of immunoglobulin (SCIg), immunoadsorption or plasma exchange within 2 weeks of the screening visit, tetracyclines with or without nicotinamide at doses higher than the recommended daily allowance (RDA)/dietary reference intake (DRI) within 2 weeks of the screening visit.
  * any monoclonal antibody (including rituximab or another anti-CD20 biologic) within 6 months of the screening visit.
  * complementary therapies-such as traditional Chinese medicines, herbs, or procedures (e.g., acupuncture)-within 4 weeks (or 5 half-lives) of the screening visit, if the investigator determines that such therapies may interfere with the study's efficacy assessments and/or potentially risk the safety of the participant.
  * The use of the following EBA treatments is permitted throughout the study: OCS, topical corticosteroids, conventional immunosuppressants (e.g., azathioprine, cyclophosphamide, methotrexate, mycophenolate, or mofetil), and dapsone.
* Moderate to severe renal insufficiency.
* Known contraindication to OCS therapy.
* Clinically significant uncontrolled active or chronic, bacterial, viral, or fungal infection at screening
* Medical instability limiting ability to travel to the Investigative Center
* Diseases or conditions that could interfere with the assessment of safety and efficacy of the study treatment and compliance of the subject with study visits/procedures, as determined by the investigator.
* Subjects actively receiving chemotherapy or immunotherapy at screening
* Active drug or alcohol addiction as determined by the investigator.
* Pregnant or nursing women
* History of malignancy unless deemed cured by adequate treatment with no evidence of recurrence for ≥3 years before the first administration of the IMP. Participants with the following cancers can be included at any time, provided they are adequately treated prior to screening:

  1. Basal cell or squamous cell skin cancer
  2. Carcinoma in situ of the cervix
  3. Carcinoma in situ of the breast
  4. Incidental histological finding of prostate cancer (TNM stage T1a or T1b)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Reduction in serum C7 antibody levels | 26 weeks
  The proportion of patients who exhibit reduction in serum C7 antibody levels at week 26 as compared to week 1.
Adverse Events and Effects | 38 weeks
  Occurrence of adverse events and effects.
EBDASI improvement | 26 weeks
  The overall improvement of EB symptoms at week 26 as compared to week 1, measured by percentage change of a participant's EBDASI score (overall total score, total activity score, and total damage score).

CONTACTS AND LOCATIONS:
Overall Officials: Matt P Marinkovich, MD, Principal Investigator — Associate Professor of Dermatology
Locations (1):
- Stanford University, Redwood City, California, United States